CLINICAL TRIAL: NCT01525680
Title: Improving PTSD Outcomes in OIF/OEF Returnees: A Randomized Clinical Trial of Hydrocortisone Augmentation of Prolonged Exposure Therapy"
Brief Title: A Randomized Clinical Trial of Hydrocortisone Augmentation of Prolonged Exposure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rachel Yehuda, MHPCCD, Bronx VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YEH-09-087
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Exposure therapy with Hydrocortisone (Active Comparator)
  Interventions: Other: Hydrocortisone augmented Prolonged Exposure Therapy
- Prolonged Exposure therapy with placebo (Placebo Comparator)
  Interventions: Other: Prolonged exposure therapy with placebo administration

INTERVENTIONS:
Other: Hydrocortisone augmented Prolonged Exposure Therapy — 11 sessions of PE. 20 minutes prior to final eight sessions, 30 mg hydrocortisone is administered.
  Arms: Prolonged Exposure therapy with Hydrocortisone
Other: Prolonged exposure therapy with placebo administration — 11 sessions of PE. 20 minutes prior to final eight sessions, placebo is administered.
  Arms: Prolonged Exposure therapy with placebo

SUMMARY:
This study seeks to examine the efficacy of hydrocortisone administration in the augmentation of the therapeutic effects of Prolonged Exposure (PE) therapy, an empirically tested treatment shown to be effective in the the treatment of posttraumatic stress disorder (PTSD). The augmentation builds on both the translation of neuroscience findings demonstrating the effects of glucocorticoids (GCs) on learning, and on empirical clinical findings from other investigators demonstrating beneficial effects of GCs in reducing traumatic memories in trauma-exposed persons.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 89
* Capable of understanding, reading, and writing in English
* OIF/OEF veteran with criterion-A trauma while deployed
* Minimum PTSD severity of 60 (CAPS)
* Unmedicated or on a stable psychotropic regimen (i.e., 1 or more months on the same regimen)

Exclusion Criteria:

* Lifetime history of psychotropic disorder, bipolar disorder, or obsessive compulsive disorder
* Moderate or severe traumatic brain injury (TBI)
* A medical or mental health problem other than PTSD that requires immediate clinical attention
* Substance abuse or dependence within the last 3 months
* Suicidal risk (as determined by response of 5 or 6 on the suicidality items of the Montgomery-Asberg Depression Rating Scale (MADRS)) and/or assessed suicide risk on the basis of clinical judgment
* Persons on a psychotropic medication regimen that has not been consistent for one month
* Presence of diabetes mellitus or any current unstable medical illness or condition that represents a contraindication to taking glucocorticoids (this will be determined by history and/or abnormal laboratory findings at medical clearance)
* Unwillingness to discontinue other specialized psychotherapy for PTSD during the 11 weeks of study treatment and the 3 month follow-up (Self-help (non-trauma focused) groups or supportive counseling can be continued but not initiated)
* Pregnant women or those planning to become pregnant within the study period will not be enrolled. Female participants must agree to use an effective method of birth control (i.e., oral contraceptive, Norplant, diaphragm, condom, or spermicide, abstinence) during the course of the study to ensure they do not become pregnant during the course of the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-04; Primary Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | week 0
  Assessment of the severity of PTSD symptoms and of diagnosis of PTSD.
Clinician Administered PTSD Scale (CAPS) | week 12
  Assessment of the severity of PTSD symptoms and of diagnosis of PTSD.
Clinician Administered PTSD Scale (CAPS) | week 23
  Assessment of the severity of PTSD symptoms and of diagnosis of PTSD.

SECONDARY OUTCOMES:
Biological measures associated with PTSD | week 0
  Measures of neuroendocrinology, genotyping, gene expression, and methylation at glucocorticoid receptor.
Biological measures associated with PTSD | week 12
  Measures of neuroendocrinology, genotyping, gene expression, and methylation at glucocorticoid receptor.
Biological measures associated with PTSD | week 23
  Measures of neuroendocrinology, genotyping, gene expression, and methylation at glucocorticoid receptor.
MATRICS Consensus Cognitive Battery (MCCB) | week 0
  Measure of cognitive ability in the following domains: processing speed, attention, working memory (verbal and non-verbal), verbal learning, visual learning, reasoning and problem solving, and social cognition.
MATRICS Consensus Cognitive Battery (MCCB) | week 12
  Measure of cognitive ability in the following domains: processing speed, attention, working memory (verbal and non-verbal), verbal learning, visual learning, reasoning and problem solving, and social cognition.
MATRICS Consensus Cognitive Battery (MCCB) | week 23
  Measure of cognitive ability in the following domains: processing speed, attention, working memory (verbal and non-verbal), verbal learning, visual learning, reasoning and problem solving, and social cognition.
Other measures of clinical, psychological, and functional outcome | week 0
  Measures of symptom severity, trauma-related cognitions, and resiliency.
Other measures of clinical, psychological, and functional outcome | week 12
  Measures of symptom severity, trauma-related cognitions, and resiliency.
Other measures of clinical, psychological, and functional outcome | week 23
  Measures of symptom severity, trauma-related cognitions, and resiliency.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Yehuda, PhD, Principal Investigator — James J Peters VAMC/Mount Sinai School of Medicine
Locations (1):
- James J. Peters Veterans Affairs Medical Center, The Bronx, New York, United States